CLINICAL TRIAL: NCT00663767
Title: A Randomized, Double-blind, Placebo- and Active-controlled, Parallel-group Analgesic Efficacy Trial of Oral ARRY-371797 in Subjects Undergoing Third Molar Extraction
Brief Title: A Study of ARRY-371797 in Subjects Undergoing Third Molar Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARRAY-797-222; C4411009 (Other: Alias Study Number)
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Dental Pain
MeSH Terms: conditions — Toothache | interventions — ARRY-371797; Celecoxib; Cyclooxygenase 2 Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; oral
- Placebo, ARRY-371797 (Experimental)
  Interventions: Drug: Placebo; oral; Drug: ARRY-371797, p38 inhibitor; oral
- ARRY-371797, Placebo (Experimental)
  Interventions: Drug: ARRY-371797, p38 inhibitor; oral; Drug: Placebo; oral
- ARRY-371797 (Experimental)
  Interventions: Drug: ARRY-371797, p38 inhibitor; oral
- Celecoxib, Placebo (Active Comparator)
  Interventions: Drug: Celecoxib, COX-2 inhibitor; oral; Drug: Placebo; oral
- Celecoxib, ARRY-371797 (Experimental)
  Interventions: Drug: Celecoxib, COX-2 inhibitor; oral; Drug: ARRY-371797, p38 inhibitor; oral

INTERVENTIONS:
Drug: Placebo; oral — dose 1, dose 2
  Arms: Placebo
Drug: Placebo; oral — dose 1
  Arms: Placebo, ARRY-371797
Drug: ARRY-371797, p38 inhibitor; oral — dose 1: multiple dose levels
  Arms: ARRY-371797, Placebo
Drug: ARRY-371797, p38 inhibitor; oral — dose 1: multiple dose levels; dose 2
  Arms: ARRY-371797
Drug: Celecoxib, COX-2 inhibitor; oral — dose 1
  Arms: Celecoxib, ARRY-371797; Celecoxib, Placebo
Drug: Placebo; oral — dose 2
  Arms: ARRY-371797, Placebo; Celecoxib, Placebo
Drug: ARRY-371797, p38 inhibitor; oral — dose 2
  Arms: Celecoxib, ARRY-371797; Placebo, ARRY-371797

SUMMARY:
This is a Phase 2 study designed to test the ability of investigational study drug ARRY-371797 to reduce pain in a postoperative pain model (third molar extraction), and to further evaluate the drug's safety. Approximately 250 subjects from the US will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Scheduled for outpatient oral surgical procedure to remove 3 or more third molars, at least 1 of which is mandibular and fully or partially impacted by bone.
* Females of childbearing potential must be willing to use an acceptable method of contraception within 14 days prior to first dose of study drug until the completion of the follow-up procedures.
* Body weight >50 kg (110 lbs).
* Good health determined by medical history, physical examination, vital signs and clinical laboratory results of non-clinical significance.
* Additional criteria exist.

Key Exclusion Criteria:

* Evidence or history of clinically significant dermatologic, hematological, renal, endocrine (e.g. poorly controlled diabetes), pulmonary, gastrointestinal, cardiovascular, hepatic, neurologic, ophthalmologic, or allergic disease (including clinically significant drug allergies that could impact the conduct of this study, but excluding untreated, asymptomatic, seasonal allergies at time of study drug dosing).
* Positive urine drug screen within 28 days prior to first dose of study drug.
* Use of prohibited prescription drugs, or grapefruit juice within 7 days of first dose of study drug; prohibited medications are defined as nonsteroidal and steroidal antiinflammatory drugs, analgesics including opioids (except low dose aspirin for myocardial infarction prophylaxis), P450 CYP3A substrates or inhibitors (strong or moderate).
* Additional criteria exist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2008-04-07 (Actual); Primary Completion 2008-06-20 (Actual); Study Completion 2008-06-20 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of the study drug dosed postoperatively in terms of total pain relief (TOTPAR). | 6 hours post-dose
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests, electrocardiograms and vital signs. | Duration of study

SECONDARY OUTCOMES:
Assess the efficacy of the study drug (versus placebo and celecoxib) in terms of pain relief measurements [including TOTPAR, total pain intensity (TPI) and time to rescue medication]. | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - PPD Phase I Clinic, Austin, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests